CLINICAL TRIAL: NCT02622880
Title: Comparison of Two Immunomodulatory Formulas on the Number of Postoperative Infections in Oropharyngeal and Maxillofacial Cancer Patients Eligible Surgery
Brief Title: Comparison of Two Immunomodulatory Formulas on the Number of Postoperative Infections in Head & Neck Cancer Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Vegenat, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VEGENAT
Record Dates: First submitted 2015-11-24; First posted 2015-12-07 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- : IMPACT (Active Comparator): along 10 days before surgery
  Interventions: Dietary Supplement: IMPACT
- immunomodulatory supplement (Experimental): along 10 days before surgery
  Interventions: Dietary Supplement: immunomodulatory supplement

INTERVENTIONS:
Dietary Supplement: immunomodulatory supplement — Experimental Group (immunomodulatory supplement STUDY)
  Arms: immunomodulatory supplement
Dietary Supplement: IMPACT — IMPACT (Nestle Healthcare Nutrition, Minnesota USA) an 'immune-enhancing' feed which contains supplemental L-arginine (1.25 78 g/L), dietary nucleotides (1.2 g/L) and omega-3 fatty acids in the form of 79 eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) (EPA/DHA 1.7 g/L) 80 as its active ingredients.
  Arms: : IMPACT

SUMMARY:
The purpose of this study is to evaluate the effect of an immune formula , consumed 10 days before surgery , on the number and characteristics of postoperative infections for a period of 30 days in a group of oropharynx, hypopharynx , larynx and oral cavity squamous cell cancer patients, candidates for surgery.

DETAILED DESCRIPTION:
68 subjects randomized into two study groups: 34 subjects consume the supplement of the study and 34 control consume the supplement IMPACT.

Intervention period will be 10 days before surgery . The consume amount is 400 ml/ day. The Subjects were stratified according to tumor location ( larynx and oral cavity and oropharynx, hypopharynx) and disease stage (early and advanced).

ELIGIBILITY:
Inclusion Criteria:

* Men and women >18 years
* Patients with histologically confirmed squamous cell cancer of the oropharynx, hypopharynx , larynx and oral cavity and candidates for neoplastic surgery (undergoing surgery)
* Adequate cultural level and understanding for the clinical trial. and agree to participate voluntarily in the study and give written informed consent
* Patients who do not participate in other clinical trials

Exclusion Criteria:

* Patients with an active infectious process at the time of the study.
* Patients who have undergone radiotherapy / chemotherapy prior to surgery.
* Subjects diagnosed with Type I Diabetes Mellitus
* Subjects who used oral hypoglycemic agents or insulin.
* Patients with severe kidney disease, heart, respiratory or liver.
* Patients with autoimmune diseases or immunosuppressive drugs used.
* Subjects with dementia, mental illness or diminished cognitive function.
* Subjects who refuse oral supplements.
* Subjects who consume vitamin supplements or artificial nutrition, and which can not be suspended at least 1 week before the study and do not accept to suspend it during the study.
* Subjects with morbid obesity (BMI ≥ 40 kg / m2).
* Pregnant or breastfeeding
* Patients diagnosed with epidermoid carcinoma T1 glottic, cordectomy candidate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Number of postoperative infections | 30 days after surgery

SECONDARY OUTCOMES:
Change from baseline Retinol-binding protein | 0 and 30 days
Length of post-operative hospital stay | through study completion, an average of 3 months
Mortality | through study completion, an average of 3 months
change from baseline C-reactive protein | 0 and 30 days
change from baseline albumin | 0 and 30 days
change from baseline transferrin | 0 and 30 days
change from baseline prealbumin | 0 and 30 days
change from baseline Bioelectrical impedance analysis | 0 and 30 days
change from baseline leukocytes | 0 and 30 days
change from baseline Fibrinogen | 0 and 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Gomez Candela, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- Hospital Universitairo La Paz, Madrid, Madrid, Spain